CLINICAL TRIAL: NCT03238391
Title: Ischemic Preconditioning for Prevention of Contrast Nephropathy in The Emergency Department: Randomised, Double Blind Clinical Trial
Brief Title: Ischemic Preconditioning for Prevention of Contrast Nephropathy in The Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Yavuz Yiğit, Emergency medicine specialist, Derince Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: kügokaek2017/51
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-07

CONDITIONS: Contrast-induced Nephropathy
Keywords: Contrast-induced nephropathy; Ischemic preconditioning
MeSH Terms: interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients will receive ischemia and reperfusion of the arm by inflating a blood pressure cuff around the arm at 50 mmHg above the systolic blood pressure for 5 minutes, followed by 5 minutes of reperfusion and this cycle will be repeated three times
  Interventions: Procedure: Ischemic preconditioning
- Sham group (Sham Comparator): Patients will receive ischemia and reperfusion of the arm by inflating a blood pressure cuff around the arm at 10 mmHg below the diastolic blood pressure for 5 minutes, followed by 5 minutes of reperfusion and this cycle will be repeated three times
  Interventions: Procedure: Ischemic preconditioning

INTERVENTIONS:
Procedure: Ischemic preconditioning — It is mentioned before in arm/group descriptions

SUMMARY:
The purpose of this study is to demonstrate the effectiveness of ischemic preconditioning in the emergency department to prevent contrast induced nephropathy

DETAILED DESCRIPTION:
The research will be conducted of emergency medicine department in The Derince Training and Research Hospital. Patients ages 18 and older, who will be received contrast enhanced CT scan in the emergency medicine department will be included to the study. Patients will be excluded from the study if The Mehran Risk Score is under 6 points. The Mehran Risk Score is a scoring system for prediction of contrast-induced nephropathy. This CIN (Contrast induced nephropathy) risk stratification score based on 8 variables. The variables included in the CIN risk score are: 1) patient-related characteristics (i.e., age >75 years, diabetes mellitus, chronic congestive heart failure, or admission with acute pulmonary edema, hypotension, anemia, and chronic kidney disease); and 2) procedure related characteristics (i.e., the use of elective IABP (Intra aortic balloon pump) or increasing volumes of contrast media). It is categorized into 4 groups according to MRS (Mehran Risk Score) (low-risk: 5 (7.5%); medium-risk: 6-10 (14%); high-risk: 11-16 (26.1%); and very high-risk: 16 (57.3%).Normal salin at a rate of 3 mL/kg/hour per 1 hour before contrast agents exposure followed by 1 mL/kg/hour for 6 hours after the procedure is administered whose Mehran risk score is greater than 6 in our daily practice. Patients with risk factors for CIN are recommended about the necessity of follow-up care with their physicians within 48-72 hours. Patients with low risk of contrast induced nephropathy, previous allergic reactions to contrast material, hemodynamically unstable and require excessive fluid resuscitation, undergoing surgical procedures, require renal-replacement therapy, who refuse to participate the study will be excluded. All of the emergency medicine physicians will be informed of the study. Participants were randomly assigned into two groups with a 1:1 allocation following simple randomization procedures by a program (www.randomization.com) generating an online random number. All participating patients will receive the standard hydration schedule as mentioned before. Patients in the study group will receive ischemia and reperfusion of the arm by inflating a blood pressure cuff around the arm at 50 mmHg above the systolic blood pressure for 5 minutes, followed by 5 minutes of reperfusion and this cycle will be repeated three times. Patients in sham group, will receive ischemia and reperfusion of the arm by inflating a blood pressure cuff around the arm at 10 mmHg below the diastolic blood pressure for 5 minutes, followed by 5 minutes of reperfusion and this cycle will be repeated three times. The allocation sequence will be concealed from the researchers and participants in sealed, sequentially numbered envelopes. Envelopes will be opened by the nurse who will administer the protocol. Less than 100 mL of nonionic, hypoosmolar contrast agent will be injected in all CT scans.All of the participants will be recommended about the necessity of follow-up care with their physicians within 48-72 hours. Participants will be called 72 hours after the treatment. Patients who are diagnosed with CIN will be followed for one month to see whether they will develop renal failure requiring renal replacement therapy. After 72 hours the laboratory results will be recorded by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Participants, older than 18 years old and received contrast enhanced CT scan in the emergency medicine department
* The Mehran Risk Score is greater than 5 points

Exclusion Criteria:

* The Mehran Risk Score is under 6 points
* Participants who doesn't want to enroll the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2017-08-15 (Estimated); Primary Completion 2018-02-15 (Estimated); Study Completion 2018-02-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants developing contrast-induced nephropathy | 48 to 72 hours
  %25 increase or a greater than 0,5 mg/dl increase in the serum creatinine level, 48 to 72 hours after the administration of contrast agent compared with the baseline creatinine measurement

SECONDARY OUTCOMES:
renal replacement theraphy | 1 month
  renal failure necessitating renal replacement therapy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Habeb M, Agac MT, Aliyev F, Pehlivanoglu S, Ongen Z. [Contrast media-induced nephropathy: clinical burden and current attempts for prevention]. Anadolu Kardiyol Derg. 2005 Jun;5(2):124-9. Turkish. PMID 15939688
- [Background] McCullough PA, Choi JP, Feghali GA, Schussler JM, Stoler RM, Vallabahn RC, Mehta A. Contrast-Induced Acute Kidney Injury. J Am Coll Cardiol. 2016 Sep 27;68(13):1465-1473. doi: 10.1016/j.jacc.2016.05.099. PMID 27659469
- [Background] Kelly AM, Dwamena B, Cronin P, Bernstein SJ, Carlos RC. Meta-analysis: effectiveness of drugs for preventing contrast-induced nephropathy. Ann Intern Med. 2008 Feb 19;148(4):284-94. doi: 10.7326/0003-4819-148-4-200802190-00007. PMID 18283206
- [Background] Marenzi G, Bartorelli AL. Recent advances in the prevention of radiocontrast-induced nephropathy. Curr Opin Crit Care. 2004 Dec;10(6):505-9. doi: 10.1097/01.ccx.0000145098.13199.e8. PMID 15616393
- [Background] Barreto R. Prevention of contrast-induced nephropathy: the rational use of sodium bicarbonate. Nephrol Nurs J. 2007 Jul-Aug;34(4):417-21. PMID 17891910
- [Background] Asif A, Garces G, Preston RA, Roth D. Current trials of interventions to prevent radiocontrast-induced nephropathy. Am J Ther. 2005 Mar-Apr;12(2):127-32. doi: 10.1097/01.mjt.0000143694.60662.11. PMID 15767830
- [Background] Ozcan EE, Guneri S, Akdeniz B, Akyildiz IZ, Senaslan O, Baris N, Aslan O, Badak O. Sodium bicarbonate, N-acetylcysteine, and saline for prevention of radiocontrast-induced nephropathy. A comparison of 3 regimens for protecting contrast-induced nephropathy in patients undergoing coronary procedures. A single-center prospective controlled trial. Am Heart J. 2007 Sep;154(3):539-44. doi: 10.1016/j.ahj.2007.05.012. PMID 17719303
- [Background] Cheung MM, Kharbanda RK, Konstantinov IE, Shimizu M, Frndova H, Li J, Holtby HM, Cox PN, Smallhorn JF, Van Arsdell GS, Redington AN. Randomized controlled trial of the effects of remote ischemic preconditioning on children undergoing cardiac surgery: first clinical application in humans. J Am Coll Cardiol. 2006 Jun 6;47(11):2277-82. doi: 10.1016/j.jacc.2006.01.066. Epub 2006 May 15. PMID 16750696
- [Background] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Background] Kharbanda RK, Li J, Konstantinov IE, Cheung MM, White PA, Frndova H, Stokoe J, Cox P, Vogel M, Van Arsdell G, MacAllister R, Redington AN. Remote ischaemic preconditioning protects against cardiopulmonary bypass-induced tissue injury: a preclinical study. Heart. 2006 Oct;92(10):1506-11. doi: 10.1136/hrt.2004.042366. Epub 2006 Jul 3. PMID 16818489
- [Background] Ali ZA, Callaghan CJ, Lim E, Ali AA, Nouraei SA, Akthar AM, Boyle JR, Varty K, Kharbanda RK, Dutka DP, Gaunt ME. Remote ischemic preconditioning reduces myocardial and renal injury after elective abdominal aortic aneurysm repair: a randomized controlled trial. Circulation. 2007 Sep 11;116(11 Suppl):I98-105. doi: 10.1161/circulationaha.106.679167. PMID 17846333
- [Background] Venugopal V, Laing CM, Ludman A, Yellon DM, Hausenloy D. Effect of remote ischemic preconditioning on acute kidney injury in nondiabetic patients undergoing coronary artery bypass graft surgery: a secondary analysis of 2 small randomized trials. Am J Kidney Dis. 2010 Dec;56(6):1043-9. doi: 10.1053/j.ajkd.2010.07.014. Epub 2010 Oct 25. PMID 20974511